CLINICAL TRIAL: NCT01659060
Title: Assessment of Blood Pressure and Endothelial Function Pregnancy After Acute and Daily Consumption Flavanol-rich Chocolate Among Healthy Pregnant Women: a Pilot Randomized Controlled Trial
Brief Title: Chocolate Consumption in Healthy Pregnant Women Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 119.05.03
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension Pregnancy-induced
Keywords: Cacao; Chocolate; Theobromine; Flavonoids; Pregnant women; Hypertension pregnancy-induced; Pre-eclampsia; Epicatechin
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dark chocolate (Experimental)
  Interventions: Other: Flavanol-rich dark chocolate
- Placebo chocolate (Placebo Comparator)
  Interventions: Other: Placebo Chocolate

INTERVENTIONS:
Other: Flavanol-rich dark chocolate — The primary objective of this pilot RCT is to test the feasibility of design methods and procedures for later use on a larger scale. The secondary objective is to examine the acute and chronic effect of dark chocolate on endothelial function and blood pressure, among healthy pregnant women.
  Other Names: Chocolate rich in flavanols
  Arms: Dark chocolate
Other: Placebo Chocolate — Placebo intervention
  Other Names: Flavanol-free chocolate
  Arms: Placebo chocolate

SUMMARY:
The purpose of this study is to to test the feasibility of design methods and procedures for later use on a larger scale and to examine the acute and chronic effect of consumption of flavanol-rich chocolate on endothelium function and blood pressure in healthy pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking normotensive women aged from 18 to 35 years, between the 7 and 12 weeks of gestation (documented by ultrasound) and having a live fetus confirmed by fetal heart auscultation

Exclusion Criteria:

* Patients with family history of premature cardiovascular disease
* Chronic hypertension
* Currently or previously use of medications interfering with glucose or lipids metabolism.
* Use of supplements or natural health products that interfere with blood pressure.
* Consumption of 1 or more alcohol drink per day.
* Allergy or intolerance to nuts or chocolate.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial function and blood pressure | within the first 12 weeks of chocolate intake (week 12 and baseline)

SECONDARY OUTCOMES:
Changes from baseline in plasma flavanol and methylxanthines(caffeine, theobromine and theophylline) concentrations at 12 weeks | within the first 12 weeks of chocolate intake (week 12 and baseline)
Weight change from baseline at 12 weeks | within the first 12 weeks of chocolate intake (week 12 and baseline)
Number of participants with digestive and other signs and symptoms (nausea, abdominal pain, constipation, and headache) | within the first 12 weeks of chocolate intake (week 12 and baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Dodin, MD, Principal Investigator — Laval University
Locations (1):
- Laval University, Department of Medicine, Institut des nutraceutiques et des aliments fonctionnels, Québec, Quebec, Canada

REFERENCES:
- [Derived] Mogollon JA, Bujold E, Lemieux S, Bourdages M, Blanchet C, Bazinet L, Couillard C, Noel M, Dodin S. Blood pressure and endothelial function in healthy, pregnant women after acute and daily consumption of flavanol-rich chocolate: a pilot, randomized controlled trial. Nutr J. 2013 Apr 8;12:41. doi: 10.1186/1475-2891-12-41. PMID 23565841